CLINICAL TRIAL: NCT02002598
Title: Phase I/II Study of Carfilzomib in Combination With Bendamustine and Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Carfilzomib With Bendamustine and Dexamethasone in Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual and loss of funding
Sponsor: Suzanne Lentzsch, MD (Other)
Responsible Party: Sponsor-Investigator, Suzanne Lentzsch, MD, Professor of Clinical Medicine, Dept of Medical Hematology & Oncology, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAJ2359
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Multiple Myeloma
Keywords: Newly diagnosed; multiple myeloma; myeloma; bendamustine; Treanda; carfilzomib; dexamethasone; phase I; phase II; dose escalation; transplant; non-transplant; plasma cell; Kyprolis
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bendamustine Hydrochloride; carfilzomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CFZ with bendamustine and dexamethasone (Experimental): Subjects will receive Carfilzomib on Days 1, 2, 8, 9, 15, and 16 every 28 days with dose escalation from 27, 36, 45 to 56 mg/ m2 . No matter what target dose the subject will receive, days 1 and 2 doses in the first cycle will always be 20 mg/m2, followed by target dose for all subsequent dates and cycles. Bendamustine will be given IV on days 1 and 2 with dose escalation up to 90 mg/m2 and dexamethasone 20 mg orally or intravenously on 1, 2, 8, 9, 15, 16, 22 and 23 of each 28-day cycle. Study treatment will be given until 8 cycles of treatment are completed or until disease progression, whichever comes first.
  Interventions: Drug: Bendamustine; Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bendamustine — Bendamustine will be administered IV on days 1 and 2 with dose escalation up to 90 mg/m2 of each 28-day cycle.
  Dose escalation is as follows:
  -1 | 60 mg/m2
  1. | 70 mg/m2
  2. | 70 mg/m2
  3. | 90 mg/m2
  4. | 90mg/m2
  5. | 90 mg/m2
  Other Names: Treanda
Drug: Carfilzomib — Carfilzomib will be administered IV on Days 1, 2, 8, 9, 15, and 16 every 28 days.
  Dose Escalation is as follows:
  -1 | 27 mg/m2
  1. | 27 mg/m2
  2. | 36 mg/m2
  3. | 36 mg/m2
  4. | 45 mg/m2
  5. | 56 mg/m2
  Other Names: Kyprolis; CFZ
Drug: Dexamethasone — Dexamethasone will be administered PO or IV, 20 mg, on 1, 2, 8, 9, 15, 16 and 22, 23 of each 28-day cycle.
  Other Names: Decadron; Dexamethasone Intensol; Dexpak Taperpak

SUMMARY:
This study is designed to define dose-limiting toxicity and determine preliminary evidence of efficacy of carfilzomib (CFZ) in combination with bendamustine and dexamethasone for patients with newly diagnosed multiple myeloma (MM).

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a malignant plasma cell disorder resulting in approximately 11,000 deaths in the United States each year. It is estimated that between 60,000-80,000 people are currently under treatment for refractory or relapsed MM. Prognosis and survival have improved over the last 20 years, but the disease is still universally fatal despite efforts to develop new and more effective chemotherapeutic regimens. Therefore, new regimens need to be developed for patients prior to peripheral blood stem cell transplant and for those unable to tolerate the toxicity of transplant.

An IRB-approved long-term retrospective chart review study (IRB-AAAU4389) was conducted to collect data for Outcome Measures relating to long-term analysis (up to 6.5 years).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Life expectancy ≥ 3 months.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
4. Adequate hepatic function.
5. Sufficient Absolute neutrophil count (ANC) within 14 days prior to randomization.
6. Sufficient Hemoglobin within 14 days prior to randomization (subjects may be receiving red blood cell (RBC) transfusions in accordance with institutional guidelines).
7. Sufficient platelet count 14 days prior to randomization.
8. Creatinine Clearance ≥ 30 mL/minute within 7 days prior to randomization.
9. Left Ventricular Ejection Fraction ≥ 40%.
10. Written informed consent in accordance with federal, local, and institutional guidelines.
11. Females of childbearing potential (FCBP) must agree to ongoing pregnancy testing and to practice contraception.
12. Male subjects must agree to practice contraception.
13. Patients must have histologically or cytologically confirmed symptomatic multiple myeloma (MM). Patients should not have previously been treated.
14. Prior kyphoplasty, vertebroplasty, local radiation therapy for symptomatic bone lesions (e.g., uncontrolled pain or high risk of pathologic fracture) are permitted.
15. Patients are allowed up to two cycles of high dose steroids if needed for symptomatic disease before study enrollment.

Exclusion Criteria:

1. Patients who have had chemotherapy for Multiple Myeloma. Exception: local radiation therapy for symptomatic bone lesions (e.g., uncontrolled pain or high risk of pathologic fracture).
2. Patients currently receiving high dose systemic steroids for treatment of Multiple Myeloma in excess of 320mg total dose of dexamethasone or equivalent, patients who received an investigational agent within 5 half-lives of the agent.
3. Patients with non-measurable Multiple Myeloma or primary plasma cell leukemia.
4. Pregnant or lactating females.
5. Major surgery within 21 days prior to enrollment.
6. Acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to enrollment.
7. Known human immunodeficiency virus (HIV) infection.
8. Known active hepatitis B or C infection.
9. Unstable angina or myocardial infarction within 4 months prior to enrollment.
10. Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to enrollment.
11. Uncontrolled, non-hematologic malignancy requiring active treatment.
12. Patients with known brain metastases (treated or not) will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
13. Significant neuropathy within 14 days prior to randomization.
14. Known history of allergy to Captisol, or to other agents in the study.
15. Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment.
16. Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to enrollment.
17. Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-11; Primary Completion 2019-03-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Lentzsch, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 23 participants signed a consent form; 2 were screen fails and 1 was removed from the study prior to the study start and did not receive the study interventions.
Groups:
- Carfilzomib 27 mg/m^2, Bendamustine 70 mg/m^2, Dexamethasone 20 mg: Participants will receive 27 mg/m^2 of Carfilzomib on Days 1, 2, 8, 9, 15, & 16 and 70 mg/m^2 of Bendamustine by IV on days 1 & 2 in a 28-day cycle. Study treatment will be given until 8 cycles of treatment are completed or until disease progression, whichever comes first. 20 mg Dexamethasone will be administered by PO or IV on Days 1, 2, 8, 9, 15, 16, 22, & 23 of each 28-day cycle.
- Carfilzomib 36 mg/m^2, Bendamustine 70 mg/m^2, Dexamethasone 20 mg: Participants will receive 36 mg/m^2 of Carfilzomib on Days 1, 2, 8, 9, 15, & 16 and 70 mg/m^2 of Bendamustine by IV on days 1 & 2 in a 28-day cycle. Study treatment will be given until 8 cycles of treatment are completed or until disease progression, whichever comes first. 20 mg Dexamethasone will be administered by PO or IV on Days 1, 2, 8, 9, 15, 16, 22, & 23 of each 28-day cycle.
- Carfilzomib 36 mg/m^2, Bendamustine 90 mg/m^2, Dexamethasone 20 mg: Participants will receive 36 mg/m^2 of Carfilzomib on Days 1, 2, 8, 9, 15, & 16 and 90 mg/m^2 of Bendamustine by IV on days 1 & 2 in a 28-day cycle. Study treatment will be given until 8 cycles of treatment are completed or until disease progression, whichever comes first. 20 mg Dexamethasone will be administered by PO or IV on Days 1, 2, 8, 9, 15, 16, 22, & 23 of each 28-day cycle.
- Carfilzomib 45 mg/m^2, Bendamustine 90 mg/m^2, Dexamethasone 20 mg: Participants will receive 45 mg/m^2 of Carfilzomib on Days 1, 2, 8, 9, 15, & 16 and 90 mg/m^2 of Bendamustine by IV on days 1 & 2 in a 28-day cycle. Study treatment will be given until 8 cycles of treatment are completed or until disease progression, whichever comes first. 20 mg Dexamethasone will be administered by PO or IV on Days 1, 2, 8, 9, 15, 16, 22, & 23 of each 28-day cycle.
- Carfilzomib 56 mg/m^2, Bendamustine 90 mg/m^2, Dexamethasone 20 mg: Participants will receive 56 mg/m^2 of Carfilzomib on Days 1, 2, 8, 9, 15, & 16 and 90 mg/m^2 of Bendamustine by IV on days 1 & 2 in a 28-day cycle. Study treatment will be given until 8 cycles of treatment are completed or until disease progression, whichever comes first. 20 mg Dexamethasone will be administered by PO or IV on Days 1, 2, 8, 9, 15, 16, 22, & 23 of each 28-day cycle.
Period: Dose Level 1
Arm/Group | Carfilzomib 27 mg/m^2, Bendamustine 70 mg/m^2, Dexamethasone 20 mg | Carfilzomib 36 mg/m^2, Bendamustine 70 mg/m^2, Dexamethasone 20 mg | Carfilzomib 36 mg/m^2, Bendamustine 90 mg/m^2, Dexamethasone 20 mg | Carfilzomib 45 mg/m^2, Bendamustine 90 mg/m^2, Dexamethasone 20 mg | Carfilzomib 56 mg/m^2, Bendamustine 90 mg/m^2, Dexamethasone 20 mg
Started | 2 | 0 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Period: Dose Level 2
Arm/Group | Carfilzomib 27 mg/m^2, Bendamustine 70 mg/m^2, Dexamethasone 20 mg | Carfilzomib 36 mg/m^2, Bendamustine 70 mg/m^2, Dexamethasone 20 mg | Carfilzomib 36 mg/m^2, Bendamustine 90 mg/m^2, Dexamethasone 20 mg | Carfilzomib 45 mg/m^2, Bendamustine 90 mg/m^2, Dexamethasone 20 mg | Carfilzomib 56 mg/m^2, Bendamustine 90 mg/m^2, Dexamethasone 20 mg
Started | 0 | 1 | 0 | 0 | 0
Completed | 0 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Dose Level 3
Arm/Group | Carfilzomib 27 mg/m^2, Bendamustine 70 mg/m^2, Dexamethasone 20 mg | Carfilzomib 36 mg/m^2, Bendamustine 70 mg/m^2, Dexamethasone 20 mg | Carfilzomib 36 mg/m^2, Bendamustine 90 mg/m^2, Dexamethasone 20 mg | Carfilzomib 45 mg/m^2, Bendamustine 90 mg/m^2, Dexamethasone 20 mg | Carfilzomib 56 mg/m^2, Bendamustine 90 mg/m^2, Dexamethasone 20 mg
Started | 0 | 0 | 1 | 0 | 0
Completed | 0 | 0 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Dose Level 4
Arm/Group | Carfilzomib 27 mg/m^2, Bendamustine 70 mg/m^2, Dexamethasone 20 mg | Carfilzomib 36 mg/m^2, Bendamustine 70 mg/m^2, Dexamethasone 20 mg | Carfilzomib 36 mg/m^2, Bendamustine 90 mg/m^2, Dexamethasone 20 mg | Carfilzomib 45 mg/m^2, Bendamustine 90 mg/m^2, Dexamethasone 20 mg | Carfilzomib 56 mg/m^2, Bendamustine 90 mg/m^2, Dexamethasone 20 mg
Started | 0 | 0 | 0 | 1 | 0
Completed | 0 | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Dose Level 5
Arm/Group | Carfilzomib 27 mg/m^2, Bendamustine 70 mg/m^2, Dexamethasone 20 mg | Carfilzomib 36 mg/m^2, Bendamustine 70 mg/m^2, Dexamethasone 20 mg | Carfilzomib 36 mg/m^2, Bendamustine 90 mg/m^2, Dexamethasone 20 mg | Carfilzomib 45 mg/m^2, Bendamustine 90 mg/m^2, Dexamethasone 20 mg | Carfilzomib 56 mg/m^2, Bendamustine 90 mg/m^2, Dexamethasone 20 mg
Started | 0 | 0 | 0 | 0 | 15
Completed | 0 | 0 | 0 | 0 | 15
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data was collected and analyzed as one arm for this single-arm study. Additionally, presented as one arm to protect the confidentiality of the first four participants.
Groups:
- CFZ With Bendamustine and Dexamethasone: First participant received: CFZ 27mg/m^2, Bendamustine 70mg/m^2, Dexamethasone 20mg; Second participant received: CFZ 36mg/m^2, Bendamustine 70mg/m^2, Dexamethasone 20mg; Third participant received: CFZ 36mg/m^2, Bendamustine 90mg/m^2, Dexamethasone 20mg; Fourth participant received: CFZ 45mg/m^2, Bendamustine 90mg/m^2, Dexamethasone 20mg; Fifth participant and all other participants received: CFZ 56mg/m^2, Bendamustine 90mg/m^2, Dexamethasone 20mg.
  Data was collected and analyzed as one arm for this single-arm study. Additionally, presented as one arm to protect the confidentiality of the first four participants.
Arm/Group | CFZ With Bendamustine and Dexamethasone
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 65 [48 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 7
  Non-Hispanic | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Carfilzomib in Combination With Bendamustine and Dexamethasone
Description: MTD defined as the highest dose at which ≤20% of participants experience dose-limiting toxicity (DLT), to define the recommended phase II dose. DLT were evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE) of the National Cancer Institute version 4.0. An AE was considered a DLT if it occurred in cycle 1, was deemed related to study treatment, and was one of peripheral neuropathy ≥grade 2, any non-hematologic AE ≥ grade 3, neutropenia grade 4 lasting ≥7 days or with fever, thrombocytopenia grade 4 lasting ≥7 days or with bleeding, or any AE requiring a dose reduction during cycle 1 or a delay in the start of cycle 2.
Time Frame: 6 months
Population: A total of 19 out of 19 participants were analyzed when evaluating the maximum tolerated dose. Participants who received dose level 5 continued to be evaluated for dose limiting toxicities.
Measure: Number; unit: mg/m^2
Groups:
- CFZ With Bendamustine and Dexamethasone: All participants who received at least two cycles of CFZ either at 27mg/m^2, 36mg/m^2, 45 mg/m^2, or 56mg/m^2.
Arm/Group | CFZ With Bendamustine and Dexamethasone
Number analyzed (Participants) | 19
mg/m^2 | 56

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR defined as the number of participants demonstrating complete response or partial response. Complete response defined as complete disappearance of an M-protein and no evidence of MM in the bone marrow. Partial response defined as ≥50% reduction in the level of the serum monoclonal paraprotein, reduction in 24-hour M-protein either by greater than or equal to 90% or to <200 mg, ≥50% reduction in size of soft tissue plasmacytoma (by radiography or clinical examination), no increase in the number or size of lytic bone lesions.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | CFZ With Bendamustine and Dexamethasone
Number analyzed (Participants) | 19
participants | 19

3. Secondary Outcome: Time to Next Treatment (TTNT)
Description: The TTNT is measured from the date of initiation of treatment to the start date of the next treatment regimen.
Time Frame: Up to 6.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CFZ With Bendamustine and Dexamethasone
Number analyzed (Participants) | 19
months | 77.0 [36.1 to NA] — The upper limit is not applicable due an to insufficient number of participants with events.

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from start of study treatment to time of progression or death, whichever occurs first.
Time Frame: Up to 6.5 Years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CFZ With Bendamustine and Dexamethasone
Number analyzed (Participants) | 19
Months | 77 [34.5 to NA] — The upper limit is not applicable due an to insufficient number of participants with events.

5. Secondary Outcome: Time to Best Response
Description: Time to the best response recorded.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CFZ With Bendamustine and Dexamethasone
Number analyzed (Participants) | 19
Months | 10.23 [4.87 to 12.96]

6. Secondary Outcome: Overall Survival (OS) Rate
Description: The percentage of people who are still alive.
Time Frame: Up to 6.5 Years
Measure: Count of Participants; unit: Participants
Arm/Group | CFZ With Bendamustine and Dexamethasone
Number analyzed (Participants) | 19
Participants | 17

7. Secondary Outcome: Number of Adverse Events (AEs)
Description: Total number of AEs observed.
Time Frame: 30 Days Post Last Dose, Up to approximately 9 months
Measure: Number; unit: Adverse Events
Arm/Group | CFZ With Bendamustine and Dexamethasone
Number analyzed (Participants) | 20
Adverse Events | 106

ADVERSE EVENTS:
Time Frame: Serious and Other Adverse Events were monitored 30 days post last dose, up to approximately 9 months. All-Cause Mortality was assessed for up to 6.5 years.
Description: Adverse events collected by investigator assessment on day 1 of each cycle and by laboratory assessment on days 1, 8, and 15 of each cycle.
Arm/Group | CFZ With Bendamustine and Dexamethasone
All-Cause Mortality (participants affected / at risk) | 2/20
Serious Adverse Events (participants affected / at risk) | 7/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CFZ With Bendamustine and Dexamethasone (N=20)
Abdominal infection (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Gastrointestinal disorders (Gastrointestinal disorders) | 1
General disorders and administration site conditions (General disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Infections and infestations (Infections and infestations) | 2
Lung infection (Infections and infestations) | 3
Platelet count decreased (Investigations) | 1
Respiratory, thoracic and mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sepsis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | CFZ With Bendamustine and Dexamethasone (N=20)
Abdominal pain (Gastrointestinal disorders) | 4/19
Agitation (Psychiatric disorders) | 2
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 2
Anal hemorrhage (Gastrointestinal disorders) | 2
Anemia (Blood and lymphatic system disorders) | 13
Anorexia (Metabolism and nutrition disorders) | 4
Anxiety (Psychiatric disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bloating (Gastrointestinal disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bronchial infection (Infections and infestations) | 1
Cardiac Disorder (Cardiac disorders) | 1
Cataract (Eye disorders) | 2
Chills (General disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Creatinine increased (Investigations) | 7
Depression (Psychiatric disorders) | 2
Diarrhea (Gastrointestinal disorders) | 8
Dizziness (Nervous system disorders) | 5
Dry mouth (Gastrointestinal disorders) | 2
Dysgeusia (Nervous system disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Edema limbs (General disorders) | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Eye Disorder (Eye disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 6
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Floaters (Eye disorders) | 1
Flu like symptoms (General disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Gastrointestinal disorders (Gastrointestinal disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 7
Hearing impaired (Ear and labyrinth disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 2
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 1
Immune system disorder (Immune system disorders) | 9
Infections and infestation (Infections and infestations) | 6
Insomnia (Psychiatric disorders) | 3
Investigations - Other (Investigations) | 1
Libido decreased (Psychiatric disorders) | 1
Lung infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 7
Malaise (General disorders) | 1
Metabolism and nutrition disorder (Metabolism and nutrition disorders) | 1
Middle ear inflammation (Ear and labyrinth disorders) | 1
Mucosal infection (Infections and infestations) | 2
Mucositis oral (Gastrointestinal disorders) | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
Nausea (Gastrointestinal disorders) | 9
Neutrophil count decreased (Investigations) | 8
Non-cardiac chest pain (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Palpitations (Cardiac disorders) | 2
Paresthesia (Nervous system disorders) | 3
Phlebitis (Vascular disorders) | 2
Phlebitis infective (Infections and infestations) | 2
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Platelet count decreased (Investigations) | 13
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Presyncope (Nervous system disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Radiculitis (Nervous system disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Rectal hemorrhage (Gastrointestinal disorders) | 1
Renal and urinary disorder (Renal and urinary disorders) | 1
Respiratory, thoracic and mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sinusitis (Infections and infestations) | 1
Skin and subcutaneous tissue disorder (Skin and subcutaneous tissue disorders) | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Stroke (Nervous system disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 4
Tooth infection (Infections and infestations) | 1
Tremor (Nervous system disorders) | 1
Upper respiratory infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 6
Urticaria (Skin and subcutaneous tissue disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Weight gain (Investigations) | 1
Weight loss (Investigations) | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
White blood cell decreased (Investigations) | 7

LIMITATIONS AND CAVEATS:
The limitations of this study include a small sample size, failure to complete planned accrual, and lack of high cytogenetic risk patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT02002598/Prot_SAP_000.pdf